CLINICAL TRIAL: NCT04532099
Title: Clinical Comparison of Two Daily Wear Frequent Replacement Silicone Hydrogel Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLY935-C020
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2021-05

CONDITIONS: Refractive Errors; Ametropia
Keywords: Contact Lenses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: Part A is a crossover study. Part B is a single group study.
Who Masked: Participant, Investigator
Masking Description: Part A is double masked. Part B is single masked (trial subject).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- LID018869, then AOHP (Part A) (Other): Lehfilcon A contact lenses worn first, followed by senofilcon A contact lenses, as randomized. Each product will be worn bilaterally (in both eyes) for approximately 30 days, with a scheduled visit at approximately Day 15 of each wear period. Lenses will be removed nightly for cleaning and disinfection with CLEAR CARE contact lens solution.
  Interventions: Device: Lehfilcon A contact lenses; Device: Senofilcon A contact lenses; Device: Hydrogen peroxide-based cleaning and disinfecting solution
- AOHP, then LID018869 (Part A) (Other): Senofilcon A contact lenses worn first, followed by lehfilcon A contact lenses, as randomized. Each product will be worn bilaterally (in both eyes) for approximately 30 days, with a scheduled visit at approximately Day 15 of each wear period. Lenses will be removed nightly for cleaning and disinfection with CLEAR CARE contact lens solution.
  Interventions: Device: Lehfilcon A contact lenses; Device: Senofilcon A contact lenses; Device: Hydrogen peroxide-based cleaning and disinfecting solution
- Biofinity (Part B) (Active Comparator): Comfilcon A contact lenses worn bilaterally (in both eyes) for approximately 30 days, with a scheduled visit at approximately Day 15 of the wear period. Lenses will be removed nightly for cleaning and disinfection with CLEAR CARE contact lens solution.
  Interventions: Device: Comfilcon A contact lenses; Device: Hydrogen peroxide-based cleaning and disinfecting solution

INTERVENTIONS:
Device: Lehfilcon A contact lenses — Investigational soft contact lenses for daily wear worn in Part A of the study
  Other Names: LID018869
  Arms: AOHP, then LID018869 (Part A); LID018869, then AOHP (Part A)
Device: Senofilcon A contact lenses — Commercially available soft contact lenses for daily wear worn in Part A of the study
  Other Names: AOHP; ACUVUE OASYS® with HYDRACLEAR® PLUS
  Arms: AOHP, then LID018869 (Part A); LID018869, then AOHP (Part A)
Device: Comfilcon A contact lenses — Commercially available soft contact lenses for daily wear worn in Part B of the study
  Other Names: CooperVision® Biofinity®
  Arms: Biofinity (Part B)
Device: Hydrogen peroxide-based cleaning and disinfecting solution — For nightly cleaning and disinfecting of contact lenses in Part A and Part B of the study
  Other Names: CLEAR CARE®

SUMMARY:
The primary objective of this study is to evaluate the overall performance of an investigational silicone hydrogel lens when compared to ACUVUE OASYS® with HYDRACLEAR® PLUS (AOHP).

DETAILED DESCRIPTION:
Part A of this study is a randomized, double masked, crossover study comparing 2 contact lens products. The expected duration of subject participation in Part A is approximately 8 weeks with 5 scheduled visits.

Part B of this study is a non-randomized, single masked, single group study with 1 contact lens product. The expected duration of subject participation in Part B is approximately 4 weeks with 3 scheduled visits.

ELIGIBILITY:
Key Inclusion Criteria:

* Sign an approved Informed Consent Form.
* Wear spherical contact lenses in both eyes for a minimum of 5 days per week and 10 hours per day during the past 3 months.
* Willing to wear habitual spectacles for vision correction when study lenses are not worn, as needed.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Any eye condition or use of medication that contraindicates contact lens wear, as determined by the Investigator.
* History of refractive surgery or plan to have refractive surgery during the study.
* Current or history of dry eye in either eye that, in the opinion of the Investigator, would preclude contact lens wear.
* Routinely sleeps in contact lenses at least 1 night per week.
* Part A: Current wearer of ACUVUE OASYS® with HYDRACLEAR® PLUS.
* Part B: Current wearer of Biofinity family of contact lenses (comfilcon A).
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Vision Care, Study Director — Alcon Research, LLC
Locations (4):
- United States (4):
  - Alcon Investigator 6356, Longwood, Florida
  - Alcon Investigator 6565, Maitland, Florida
  - Alcon Investigator 6401, Warwick, Rhode Island
  - Alcon Investigator 6353, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 investigative sites located in the United States.
Groups:
- LID018869, Then AOHP (Part A): Lehfilcon A contact lenses worn first, followed by senofilcon A contact lenses, as randomized. Each product was worn bilaterally (in both eyes) for approximately 30 days, with a scheduled visit at approximately Day 15 of each wear period. Lenses were removed nightly for cleaning and disinfection with CLEAR CARE contact lens solution.
- AOHP, Then LID018869 (Part A): Senofilcon A contact lenses worn first, followed by lehfilcon A contact lenses, as randomized. Each product was worn bilaterally (in both eyes) for approximately 30 days, with a scheduled visit at approximately Day 15 of each wear period. Lenses were removed nightly for cleaning and disinfection with CLEAR CARE contact lens solution.
- Biofinity (Part B): Comfilcon A contact lenses worn bilaterally (in both eyes) for approximately 30 days, with a scheduled visit at approximately Day 15 of the wear period. Lenses were removed nightly for cleaning and disinfection with CLEAR CARE contact lens solution.
Period: First Wear Period (30 Days)
Arm/Group | LID018869, Then AOHP (Part A) | AOHP, Then LID018869 (Part A) | Biofinity (Part B)
Started | 33 | 33 | 66
Completed | 32 | 33 | 66
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Second Wear Period (30 Days)
Arm/Group | LID018869, Then AOHP (Part A) | AOHP, Then LID018869 (Part A) | Biofinity (Part B)
Started | 32 | 33 | 0 (Part B is single product; therefore, only one wear period.)
Completed | 32 | 33 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID018869, Then AOHP (Part A) | AOHP, Then LID018869 (Part A) | Biofinity (Part B) | Total
Number analyzed (Participants) | 33 | 33 | 66 | 132
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 33 | 33 | 66 | 132
  Equal to or greater than 65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 49 | 95
  Male | 7 | 13 | 17 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 5 | 7
  Not Hispanic or Latino | 32 | 32 | 61 | 125
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 4
  White | 31 | 32 | 62 | 125
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (VA) (Part A)
Description: Distance VA was assessed with study lenses in place. VA was collected for each eye separately using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity. No formal hypothesis testing was predefined for the primary endpoint. The primary endpoint was prespecified for Part A only.
Time Frame: Day 30, each study lens type
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID018869 (Part A): Lehfilcon A contact lenses worn during Period 1 or Period 2, as randomized, for approximately 30 days. Lenses were removed nightly for cleaning and disinfection with CLEAR CARE contact lens solution.
- AOHP (Part A): Senofilcon A contact lenses worn during Period 1 or Period 2, as randomized, for approximately 30 days. Lenses were removed nightly for cleaning and disinfection with CLEAR CARE contact lens solution.
Arm/Group | LID018869 (Part A) | AOHP (Part A)
Number analyzed (Participants) | 66 | 65
Number analyzed (eyes) | 132 | 130
logMAR | -0.12 (0.09) | -0.12 (0.09)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 8 weeks for subjects enrolled in Part A and approximately 4 weeks for subjects enrolled in Part B.
Description: An AE was defined at any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the test article. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. At Risk" population of pretreatment and non-ocular AEs is reported in units of subjects; all other AE populations are reported in units of eyes.
Groups:
- Pretreatment Part A; Pretreatment Part B: Events reported in this group occurred prior to exposure to the study contact lenses.
- LID018869 Ocular (Part A); LID018869 Nonocular: Events reported in this group occurred while exposed to lehfilcon A contact lenses.
- AOHP Ocular; AOHP Nonocular: Events reported in this group occurred while exposed to senofilcon A contact lenses.
- Biofinity Ocular; Biofinity Nonocular: Events reported in this group occurred while exposed to comfilcon A contact lenses.
Arm/Group | Pretreatment Part A | LID018869 Ocular (Part A) | LID018869 Nonocular | AOHP Ocular | AOHP Nonocular | Pretreatment Part B | Biofinity Ocular | Biofinity Nonocular
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/132 | 0/66 | 0/130 | 0/65 | 0/66 | 0/132 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/132 | 0/66 | 0/130 | 0/65 | 0/66 | 0/132 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/132 | 0/66 | 0/130 | 0/65 | 0/66 | 0/132 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT04532099/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT04532099/SAP_001.pdf